CLINICAL TRIAL: NCT05530265
Title: Effect of Smart Watch and App on Positive Airway Pressure Adherence in Patients With Obstructive Sleep Apnea: A Randomized Controlled Trial
Brief Title: Effect of Smart Watch and App on PAP Adherence in OSA (Watch-OSA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jaeyoung Cho, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22070571340
Record Dates: First submitted 2022-09-03; First posted 2022-09-07 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea of Adult; Positive Airway Pressure; Adherence, Treatment; Smart Watch
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart watch group (Experimental): The user of the smart watch and Samsung Health app
  Interventions: Device: the smart watch and Samsung Health app
- Usual care (No Intervention): No use of both the smart watch and Samsung Health app

INTERVENTIONS:
Device: the smart watch and Samsung Health app — Use the smart watch (Galaxy Watch 4, Samsung Electronics Co., Ltd., Korea) and the Samsung Health app (Samsung Electronics Co., Ltd., Korea) for 90 days of positive airway pressure treatment
  Arms: Smart watch group

SUMMARY:
Continuous positive airway pressure (CPAP) is highly effective in treating obstructive sleep apnea (OSA). However, this treatment modality relies heavily on patient adherence, and poor adherence to the treatment limits its effectiveness in treating OSA. Strategies to augment adherence are needed in the management of OSA.

The smart watch and linked app provide various health information, including sleep, snoring or oxygen saturation during sleep, exercise, blood pressure, and electrocardiogram. The smart watch and linked app could potentially improve adherence to positive airway pressure (PAP) treatment.

This randomized controlled trial (RCT) aimed to examine whether the use of smart watch and app can increase PAP adherence in patients with OSA.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with OSA (apnea-hyponea index [AHI])≥ 5 /h) by type 1 polysomnography
* no prior use of PAP (CPAP or auto-adjusting PAP [APAP]), or no prior use of PAP within the previous 90 days in patients who had received PAP therapy, or current PAP users with average daily usage (all days) < 4 hours within the previous 90 days

Exclusion Criteria:

* patients who refuse PAP therapy
* patients who have used a smart watch (e.g., Galaxy Watch, Apple Watch, etc.) within the previous 90 days
* patients with central sleep apnea or neuromuscular disease
* patients receiving supplemental oxygen therapy due to underlying diseases including heart failure, stroke, chronic obstructive pulmonary disease, interstitial pulmonary disease, hypoventilation syndrome, or whose baseline oxygen saturation is less than 90%
* patients with implanted cardiac pacemakers, defibrillators, or other electronic devices
* patients who are inexperienced in using smartphones, apps, or smart watches
* patients with an inability or unwillingness to provide informed consent

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Average daily usage of PAP (all days) | 90 days
  Average daily usage of PAP (all days) in 90 days

SECONDARY OUTCOMES:
Average daily usage of PAP (days used) | 90 days
  Average daily usage of PAP (days used) in 90 days
Percentage of days using PAP | 90 days
  Percentage of days using PAP
Percentage of days using PAP ≥ 4 hours | 90 days
  Percentage of days using PAP ≥ 4 hours
Percentage of patients meeting the National Health Insurance Service adherence criteria | 90 days
  The National Health Insurance Service adherence criteria: ≥ 4 hours of use on ≥ 70% of days over 30 consecutive days during the 90 days of PAP therapy
Changes of the scores of Epworth Sleepiness Scale | 90 days
  Changes of the scores of Epworth Sleepiness Scale
Changes of the scores of Pittsburgh Sleep Quality Index | 90 days
  Changes of the scores of Pittsburgh Sleep Quality Index (an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality)
Patient satisfaction with PAP therapy | 90 days
  Patient satisfaction with PAP therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jaeyoung Cho, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea